CLINICAL TRIAL: NCT06326229
Title: Clinical Validation of the Content of an ICF Core Set for the Management of Musculoskeletal Conditions in Primary Care Physiotherapy Services
Brief Title: Clinical Validation of Musculoskeletal ICF Core Set in Primary Care Physiotherapy
Status: Recruiting | Type: Observational
Sponsor: University of Valladolid (Other)
Collaborators: Castilla-León Health Service (Other)
Responsible Party: Principal Investigator, Héctor Hernández Lázaro, Principal Investigator, University of Valladolid
Other Study IDs: CEIm 3096
Record Dates: First submitted 2024-03-16; First posted 2024-03-22 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Musculoskeletal Diseases
Keywords: Musculoskeletal Diseases, ICF, Primary Health Care, Physical Therapy Modalities
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Musculoskeletal patients: Patients suffering from musculoskeletal problems referred by a family physician for management in primary care physiotherapy services.
  Interventions: Other: ICF entities assessment

INTERVENTIONS:
Other: ICF entities assessment — A visual analog scale will be used by the participants to evaluate the relevance of the ICF entities in relation to their musculoskeletal condition. The scale will range from 0 (no problem) to 100 (complete problem).

SUMMARY:
The aim of this observational study is to validate the content of a tailored ICF core set for the management of musculoskeletal conditions in primary care physiotherapy services.

The main question it aims to answer is:

- Are the ICF entities included in the ICF Core Set under evaluation useful from a clinical point of view?

Participants will evaluate the relevance of each ICF entity included in the ICF core set according to their musculoskeletal condition.

DETAILED DESCRIPTION:
Primary care physiotherapy services provide community-based care for musculoskeletal conditions. These conditions are often associated with disability and impact on patients' quality of life. The International Classification of Functioning, Disability and Health (ICF) is the global framework for describing disability. ICF Core Sets are ICF-based tools that facilitate the clinical use of this classification. Some ICF Core Sets are designed to describe the functioning of patients with musculoskeletal problems.

These Core Sets are focused on the acute phase, typical of emergency care, and the post-acute phase, intended for multidisciplinary teams in rehabilitation centers. However, no ICF core set exists for the final stages of these conditions, when the patient has been reintegrated into the community. The development of ICF Core Sets follows a scientific process that integrates the perspectives of researchers, patients, professionals, and the care setting. Therefore, preparatory studies were carried out, taking as a reference the physiotherapy services in primary care, where most of these conditions are treated. A preliminary ICF core set was developed from these studies, the entities of which were agreed upon through a subsequent cross-sectional study involving a group of primary care physiotherapy experts. In order to confirm the usefulness of this ICF core set, a cross-sectional study will be developed to assess the clinical relevance of the ICF entities included in it.

A multicenter cross-sectional observational study will be carried out in primary care physiotherapy services to assess the relevance of various aspects of functioning in patients with musculoskeletal problems. The participants will be people suffering from musculoskeletal problems referred to these services for treatment by a general practitioner. The ICF core set will be used as outcome measure and the relevance of its ICF entities will be assessed by the participants. For this purpose, a 100 mm visual analog scale will be used, where 0 will mean "no problem" and 100 will mean "complete problem". Scores will be converted into ICF qualifiers. The criterion for confirming each ICF entity will be that it represents a problem in at least 5% of the sample. Confirmation of the ICF entities will allow the development of an ICF-based clinical tool for the management of musculoskeletal conditions in primary care physiotherapy services.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Patients diagnosed with a musculoskeletal condition by a general practitioner
* Patients with adequate knowledge of the Spanish language

Exclusion Criteria:

* Patients referred for a non-musculoskeletal problem
* Patients referred from hospital services

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be the group of patients referred by a general practitioner to physiotherapy services in primary care for the management of musculoskeletal problems.
Sampling Method: Non-Probability Sample
Enrollment: 385 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-09-26 (Estimated)

PRIMARY OUTCOMES:
ICF core set for post-acute musculoskeletal conditions (adapted version for primary care physiotherapy services) | 2024-05/2024-12
  The ICF entities to be used have been obtained in an observational study with registry number NCT06168721. The list of categories will be available in this registry once the study is published.

OTHER OUTCOMES:
Sociodemographic data of the sample | 2024-05/2024-12
  Data set for the characterization of the sample (age, gender, education level, job and musculoskeletal diagnosis)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Jiménez del Barrio, PhD, Study Chair — University of Valladolid; Luis Ceballos Laita, PhD, Study Chair — University of Valladolid; María Teresa Mingo Gómez, PhD, Study Chair — University of Valladolid
Locations (1):
- Ólvega Primary Care Physiotherapy service, Ólvega, Soria, Spain

IPD SHARING:
Plan to Share IPD: Yes
The authors confirm that the data supporting the findings of this study will be available within the article and/or its supplementary materials.
Supporting Information: Study Protocol, SAP
Time Frame: From the publication of the study, with no time limit.
Access Criteria: Access to this data will be conditioned by the type of publication.

REFERENCES:
- [Background] Hernandez-Lazaro H, Mingo-Gomez MT, Ceballos-Laita L, Medrano-de-la-Fuente R, Jimenez-Del Barrio S. Validation of the international classification of functioning, disability, and health (ICF) core sets for musculoskeletal conditions in a primary health care setting from physiotherapists' perspective using the Delphi method. Disabil Rehabil. 2023 Jul;45(15):2458-2468. doi: 10.1080/09638288.2022.2096128. Epub 2022 Jul 13. PMID 35830343
- [Background] Hernandez-Lazaro H, Mingo-Gomez MT, Jimenez-Del-Barrio S, Lahuerta-Martin S, Hernando-Garijo I, Medrano-de-la-Fuente R, Ceballos-Laita L. Researcher's Perspective on Musculoskeletal Conditions in Primary Care Physiotherapy Units through the International Classification of Functioning, Disability, and Health (ICF): A Scoping Review. Biomedicines. 2023 Jan 20;11(2):290. doi: 10.3390/biomedicines11020290. PMID 36830831
- [Background] Hernandez-Lazaro H, Mingo-Gomez MT, Jimenez-Del-Barrio S, Rodriguez-Fernandez AI, Areso-Boveda PB, Ceballos-Laita L. Validation of the International Classification of Functioning, Disability, and Health (ICF) core set for post-acute musculoskeletal conditions in a primary care physiotherapy setting from the perspective of patients using focus groups. Disabil Rehabil. 2024 Aug;46(16):3594-3601. doi: 10.1080/09638288.2023.2251392. Epub 2023 Sep 5. PMID 37667886
- [Background] Hernandez-Lazaro H, Jimenez-Del Barrio S, Ceballos-Laita L, Lahuerta-Martin S, Medrano-de-la-Fuente R, Hernando-Garijo I, Mingo-Gomez MT. Multicentre cross-sectional study assessing content validity of the International Classification of Functioning, disability and health core set for post-acute musculoskeletal conditions in primary care physiotherapy services. J Rehabil Med. 2023 Nov 16;55:jrm11950. doi: 10.2340/jrm.v55.11950. PMID 37974517